CLINICAL TRIAL: NCT00938678
Title: A Phase I, Randomized, Single Dose, Crossover Study Evaluating the Pharmacokinetics and Pharmacodynamics of Pegfilgrastim Hospira Compared to Neulasta (Amgen) Following Subcutaneous Administration to Healthy Volunteers
Brief Title: Pharmacokinetic/Pharmacodynamic (PK/PD) Study Evaluating Pegfilgrastim Hospira Compared to Neulasta (Amgen) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PEG-09-01; EudraCT Number 2009-101433-42
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2015-06

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group 1 (Experimental)
  Interventions: Drug: Pegfilgrastim Hospira
- Treatment Group 2 (Active Comparator)
  Interventions: Drug: Neulasta (Amgen)

INTERVENTIONS:
Drug: Pegfilgrastim Hospira — Subjects in both treatment groups will have safety assessments and will be followed for all adverse and serious adverse events.
  Arms: Treatment Group 1
Drug: Neulasta (Amgen) — Subjects in both treatment groups will have safety assessments and will be followed for all adverse and serious adverse events.
  Arms: Treatment Group 2

SUMMARY:
This study compared the pharmacokinetics, pharmacodynamics and the safety of Pegfilgrastim Hospira and Neulasta® following a single dose of 6 mg of each product administered subcutaneously in Treatment Periods 1 and 2, respectively, in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects, 18-55 years inclusive.
* Written informed consent given
* Willing and able to comply with the requirements of the protocol and be available for the planned duration of the study.
* Body Mass Index (BMI) between 19 and 30 kg/m2 inclusive and weight not <50 kg or >100 kg.
* Female subjects who are using an effective method of contraception, or are surgically sterile.
* Non-smokers or ex-smokers who have not smoked within the previous 12 months.

Exclusion Criteria:

* Hypersensitivity to the Investigational medicinal product (IMP) or its constituents and/or hypersensitivity to E. Coli derived proteins, and/or previous exposure to the IMP.
* History or presence of any clinically significant findings that, in the opinion of the Investigator, would preclude inclusion in the study.
* History or presence of any clinically significant gastrointestinal pathology or symptoms, liver or kidney disease, or any other condition that might interfere with the absorption, distribution, metabolism or excretion of the drug.
* Any clinically significant laboratory findings, including any ANC, platelet or haemoglobin result outside the reference range of the local laboratory.
* Abnormal vital signs or abnormal 12-lead electrocardiogram (ECG) results, as judged by the Investigator to be clinically significant.
* Females, pregnant or lactating, or planning to become pregnant during the time the subject is on study.
* Subjects with a history of pulmonary infiltrate or pneumonia in the previous 6 months from the date of the screening visit.
* Hereditary fructose intolerance.
* Participation in any other clinical trial using a investigational product or device, within the previous 12 weeks from the date of the screening visit.
* Positive result for human immunodeficiency virus (HIV) and/or hepatitis B and C tests.
* Evidence of, or treatment for, drug or alcohol abuse within one year from date of screening visit.
* Blood donation >=500 mL in the previous 12 weeks from the date of the screening visit.
* Use of any prescription medication (excluding hormonal contraceptives) within 14 days prior to date of the screening visit.
* Receipt of over-the-counter medicines which have not yet cleared from the body (five half-lives must have passed for the medicine to be considered to have cleared from the body). Vitamins, minerals and nutritional supplements may be taken at the discretion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time 0 extrapolated to infinity (AUC0-∞) for serum Pegfilgrastim (PEG-GCSF) | Treatment Periods 1 and 2: Pre-dose (-15 min) and post-dose 1, 2, 4, 6, 8, 10, 16, 24±2, 48±2, 72±2, 96±2, 120±2, 144±2, 168±2, 192±2, 216±2, 240±2, 264±2, 288±2 hours or early discontinuation.
Area under the curve from time 0 to the last time point (AUC0-t) for serum Pegfilgrastim (PEG-GCSF) | Treatment Periods 1 and 2: Pre-dose (-15 min) and post-dose 1, 2, 4, 6, 8, 10, 16, 24±2, 48±2, 72±2, 96±2, 120±2, 144±2, 168±2, 192±2, 216±2, 240±2, 264±2, 288±2 hours or early discontinuation.
  AUC0-t will be used as a primary parameter only if AUC0-∞ cannot be calculated for all subjects in the pharmacokinetic population.
Pharmacodynamics: Maximum change from baseline in absolute neutrophil count (ANC); ANC_Cmax | Screening, Day -1, Treatment Periods 1 & 2: Pre-dose (-60 min, -30 min, 0 min), Post dose (12 hr, 24±2, 48±2, 72±2, 96±2, 120±2, 144±2, 168±2, 192±2, 216±2, 240±2, 264±2, 288±2)

SECONDARY OUTCOMES:
Maximum concentration (Cmax) for serum Pegfilgrastim (PEG-GCSF) | Treatment Periods 1 and 2: Pre-dose (-15 min) and post-dose 1, 2, 4, 6, 8, 10, 16, 24±2, 48±2, 72±2, 96±2, 120±2, 144±2, 168±2, 192±2, 216±2, 240±2, 264±2, 288±2 hours or early discontinuation.
Time to maximum concentration (Tmax) for serum Pegfilgrastim (PEG-GCSF) | Treatment Periods 1 and 2: Pre-dose (-15 min) and post-dose 1, 2, 4, 6, 8, 10, 16, 24±2, 48±2, 72±2, 96±2, 120±2, 144±2, 168±2, 192±2, 216±2, 240±2, 264±2, 288±2 hours or early discontinuation.
Terminal elimination rate constant (λz) for serum Pegfilgrastim (PEG-GCSF) | Treatment Periods 1 and 2: Pre-dose (-15 min) and post-dose 1, 2, 4, 6, 8, 10, 16, 24±2, 48±2, 72±2, 96±2, 120±2, 144±2, 168±2, 192±2, 216±2, 240±2, 264±2, 288±2 hours or early discontinuation.
Half-life (T½) for serum Pegfilgrastim (PEG-GCSF) | Treatment Periods 1 and 2: Pre-dose (-15 min) and post-dose 1, 2, 4, 6, 8, 10, 16, 24±2, 48±2, 72±2, 96±2, 120±2, 144±2, 168±2, 192±2, 216±2, 240±2, 264±2, 288±2 hours or early discontinuation.
Area under the curve above baseline of ANC [ANC_AUC(0-tlast)] | Screening, Day -1, Treatment Periods 1 & 2: Pre-dose (-60 min, -30 min, 0 min), Post dose (12 hr, 24±2, 48±2, 72±2, 96±2, 120±2, 144±2, 168±2, 192±2, 216±2, 240±2, 264±2, 288±2)
Time of maximum change from baseline for ANC in days (ANC_Tmax) | Screening, Day -1, Treatment Periods 1 & 2: Pre-dose (-60 min, -30 min, 0 min), Post dose (12 hr, 24±2, 48±2, 72±2, 96±2, 120±2, 144±2, 168±2, 192±2, 216±2, 240±2, 264±2, 288±2)
Maximum change from baseline in CD34+ count (CD34+_Cmax) | Day -1, Treatment Periods 1 & 2: Post dose (12 hr, 24±2, 48±2, 72±2, 96±2, 120±2, 144±2, 168±2, 192±2, 216±2, 240±2)
Time of maximum change from baseline for CD34+ count in days (CD34+_Tmax) | Day -1, Treatment Periods 1 & 2: Post dose (12 hr, 24±2, 48±2, 72±2, 96±2, 120±2, 144±2, 168±2, 192±2, 216±2, 240±2)

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical Ltd, Edinburgh, United Kingdom